CLINICAL TRIAL: NCT00514787
Title: Be SMART NIS, Moderate to Servere Asthma Patient Observation
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Other Study IDs: NIS-RAT-SYM-2007/1
Record Dates: First submitted 2007-08-09; First posted 2007-08-10 (Estimated); Last update posted 2009-03-27 (Estimated); Status verified 2009-03

CONDITIONS: Asthma
Keywords: Asthma; NIS
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Screen for moderate to severe asthma patients with suboptimal asthma control (as defined by GINA-Guidelines). Document current asthma control status. Re-evaluate asthma therapy and document new therapy if applicable.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe asthma with suboptimal control

Exclusion Criteria:

* Intermittent or mild asthma, patient with good asthma control

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 900 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Pohl, PHD, Study Chair — Executive Board OGP (Austria Society of Pneumology
Locations (1):
- Research Site, Vienna, Austria